CLINICAL TRIAL: NCT04505371
Title: Improving the Reach and Effectiveness of Smoking Cessation Services Targeted to Veterans Living With HIV
Brief Title: Improving the Reach & Effectiveness of Smoking Cessation Services Targeted to Veterans Living With HIV
Acronym: WISH
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Seattle Institute for Biomedical and Clinical Research (Other)
Collaborators: Kaiser Permanente (Other); University of California, Davis (Other); Fred Hutchinson Cancer Center (Other); US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1R01CA243907-01 (NIH)
Record Dates: First submitted 2020-07-30; First posted 2020-08-10 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: HIV Infections; Smoking; Smoking Cessation
Keywords: HIV; Smoking; Smoking Cessation; Behavioral Intervention; Remote Intervention; Motivational Interviewing; Veterans
MeSH Terms: conditions — HIV Infections; Smoking; Smoking Cessation | interventions — Seroconversion

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control - Standard Care (No Intervention): The control intervention is referral to standard evidence-based cessation services available nationally to Veterans, including the National VA Quitline and SmokefreeVET texting program.
- Intervention - Wellness Intervention for Smokers with HIV (Experimental): The experimental WISH intervention is an HIV-specific comprehensive wellness program designed to offer integrated phone and text counseling regardless of readiness to quit.
  Interventions: Behavioral: Wellness Intervention for Smokers with HIV

INTERVENTIONS:
Behavioral: Wellness Intervention for Smokers with HIV — WISH is delivered remotely by mobile phone (voice and text message). WISH addresses both smoking and a number of other personally relevant health behaviors (such as treatment engagement, medication adherence, stress and mood management, social support, alcohol use, etc.), making it relevant and engaging to all, not just those ready to stop smoking. For those not yet ready to quit, WISH is designed to build and strengthen motivation and self-confidence for quitting, while smokers also work on other personal health goals.
  Once ready to quit smoking, participants receive evidence-based cognitive-behavioral counseling and encouragement to access nicotine replacement therapy (NRT) or other appropriate pharmacotherapy through usual care VA procedures. Medications will not be prescribed or dispensed by the study.
  Arms: Intervention - Wellness Intervention for Smokers with HIV

SUMMARY:
This project will compare the effectiveness of an HIV-specific comprehensive wellness intervention designed to have broad appeal to smokers living with HIV to the effectiveness of standard care services that include referral to the National VA Quitline and SmokefreeVET texting program. Participants in both arms will have access to pharmacotherapy available through their Veterans Affairs (VA) healthcare providers.

DETAILED DESCRIPTION:
Tobacco use remains the leading preventable cause of death and illness in our society, and smoking rates are disproportionately high among people living with HIV. NCI, nicotine dependence researchers, and HIV clinicians have all called for research to evaluate targeted and tailored smoking cessation programs for smokers living with HIV (SLWH). Research suggests SLWH are largely unaware of the HIV-specific deleterious effects of smoking and often lack motivation and confidence in their ability to quit. For these reasons, we developed the Wellness Intervention for Smokers with HIV (WISH).

Similar to standard care cessation services available to Veterans, WISH is delivered remotely by mobile phone (voice and text message). The program is designed for all SLWH, regardless of their initial motivation to quit. WISH follows evidence-based, best practice guidelines for nicotine dependence treatment, but is innovative in its use of a more comprehensive wellness approach. That is, the intervention addresses both smoking and a number of other personally relevant health behaviors (such as treatment engagement, medication adherence, stress and mood management, social support, alcohol use, etc.), making it relevant and engaging to all SLWH, not just those ready to stop smoking. For those not yet ready to quit, WISH is designed to build and strengthen motivation and self-confidence for quitting, while smokers also work on other personal health goals.

Once ready to quit smoking, participants receive evidence-based cognitive-behavioral counseling and encouragement to access nicotine replacement therapy (NRT) or other appropriate pharmacotherapy through usual care VA procedures. Medications will not be prescribed or dispensed by the study, allowing use of these standard services to be compared across study groups.

In this two-group randomized trial, we will compare the effectiveness of WISH to standard care services offered through the National VA Quitline and the SmokefreeVET texting program (tobacco cessation services available to all Veterans). Participants in both study groups can receive phone/ text counseling and have access to pharmacotherapy through VA. Cessation services in both study groups will be provided and overseen by the non-VA sites that developed each program.

Smoking-related outcomes will include 7-day point prevalence smoking abstinence and presence of any 24-hour intentional quit attempts, prolonged abstinence, and change in cigarettes per day. We will measure change in smoking-related knowledge, motivation and behavioral skills, as well as intervention reach and implementation. We will also describe comorbidities and explore intervention impact on markers of immune status and mortality risk using clinical data resources available through the Veterans Aging Cohort Study (VACS).

If effective, WISH could meaningfully increase the reach of cessation services and reduce smoking among HIV+ Veterans nationwide. To support this goal, dissemination efforts are planned in Year 5 to share the WISH program with the National VA Quitline. Because VA is the largest U.S. provider of HIV care, this research has the potential for significant public health impact.

ELIGIBILITY:
Inclusion Criteria:

* In care in the VA
* HIV+ serostatus
* Currently smoking 5+ cigarettes daily
* Access to cell phone with text messaging capabilities
* English speaking

Exclusion Criteria:

* Psychosis, dementia or significant cognitive impairment documented in the EHR
* Documented or observed hearing or comprehension difficulties that would preclude participation in study telephone calls
* Currently receiving cessation counseling or using an FDA approved treatment to quit smoking
* Institutionalized/imprisoned
* Pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 226 (Estimated)
Dates: Start 2021-06-04 (Actual); Primary Completion 2025-03-31 (Actual); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
7-day point-prevalence abstinence (PPA) | 6 months post-randomization
  Smoking abstinence at 6-month follow-up by self-report and biochemically confirmed via saliva cotinine for a small selected group of individuals. Cotinine levels < 10 ng/ml and a self-report of 7 day PPA will be required to be coded a nonsmoker.
Any 24-hour intentional quit attempt | 3 and 6 months postrandomization
  The primary outcome will be presence of an intentional quit attempt [yes/no] reported between randomization and 6 month follow-up. Quit attempts will be assessed at each follow-up.

SECONDARY OUTCOMES:
Floating prolonged abstinence | 3 and 6 months post-randomization
  A proxy for sustained abstinence appropriate for evaluating a motivational intervention, in which the start point floats based on one's actual quit date rather than a pre-determined quit date
7-day self-report point-prevalence abstinence (PPA) | 3 and 6 months post-randomization
  Self-report of abstinence from smoking, even a puff
30-day self-report point-prevalence abstinence (PPA) | 3, 6, 12 months post-randomization
  Self-report of abstinence from smoking, even a puff
Cigarettes smoked per day | 3 and 6 months post-randomization
  Self-report; even a puff counts as smoking
HIV-specific smoking knowledge | 3 and 6 months post-randomization
  Items validated in a survey of Smokers Living with HIV conducted by the study team during a study titled "Smoking cessation-related information, motivation, and behavioral skills specific to HIV-infected smokers" (likert scale)
Motivation to quit smoking | 3 and 6 months post-randomization
  1-10 likert scale
Smoking cessation related to self-efficacy | 3 and 6 months post-randomization
  1-10 likert scale on domains (each) of quitting smoking, reducing smoking, managing cravings, and stimulus control
Nicotine withdrawal symptom management (behavioral skills) | 3 and 6 months post-randomization
  Self-report Minnesota Smoking Withdrawal Scale, Revised
Cessation medication use and adherence (behavioral skills) | 3 and 6 months post-randomization
  Self-report and health records (pharmacy) monitoring
Absolute CD4 count | 6 and 12 months post-randomization
  Lab value of CD4 ascertained via EHR
VACS index 2.0 | 6 and 12 months post-randomization
  Composite score based of various lab values ascertained via EHR
Intentional quit attempt frequency and duration | 3 and 6 months post-randomization
  Behavioral Risk Factor Surveillance System (BRFSS)

CONTACTS AND LOCATIONS:
Overall Officials: Kristina Crothers, MD, Principal Investigator — VA Puget Sound Health Care System
Locations (1):
- VA Puget Sound Health Care System Seattle Division, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: Undecided